CLINICAL TRIAL: NCT00192842
Title: Phase II Trial of Gemcitabine and Curcumin in Patients With Advanced Pancreatic Cancer
Brief Title: Gemcitabine With Curcumin for Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RonCurcuminPancreas.CTIL
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2010-09-22 (Estimated); Status verified 2010-09

CONDITIONS: Pancreatic Cancer
Keywords: carcinoma; pancreas; gemcitabine; curcumin
MeSH Terms: conditions — Pancreatic Neoplasms; Carcinoma | interventions — Curcumin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: curcumin (+ gemcitabine)

SUMMARY:
The study hypotheasis is that curcumin, a natural compound with a potent antiproliferative effect, can improve the efficacy of the standard chemotherapy gemcitabine in patients with advanced pancreatic cancer. That is why the patients are given a daily oral dose of 8 gr of curcumin along the chemotherapeutic protocol of weekly gemcitabine.

ELIGIBILITY:
Inclusion Criteria:

* locally advanced or metastatic adenocarcinoma of the pancreas
* no prior chemotherapy
* performance status 0-2
* adequate hematology and chemistry

Exclusion Criteria:

* serious concurrent medical condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2004-07; Primary Completion 2007-11 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
time to tumor progression

SECONDARY OUTCOMES:
response rate
survival
clinical benefit
toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Ron Epelbaum, MD, Principal Investigator